CLINICAL TRIAL: NCT07120048
Title: A Prospective, Observational Registry Study Designed to Collect Real-world Hemodynamic and Clinical Outcomes of the INSPIRIS RESILIA Aortic Valve
Brief Title: Real World Data Collection on the INSPIRIS RESILIA Aortic Valve
Acronym: INDICATE
Status: Recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2025-07
Record Dates: First submitted 2025-07-31; First posted 2025-08-13 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | US Export: Yes

GROUPS / COHORTS (1):
- Edwards INSPIRIS RESILIA Aortic Valve: Subjects who were treated with the INSPIRIS RESILIA Aortic Valve
  Interventions: Device: Edwards INSPIRIS RESILIA Aortic Valve

INTERVENTIONS:
Device: Edwards INSPIRIS RESILIA Aortic Valve — Surgical replacement of the aortic valve with the Edwards INSPIRIS RESILIA Aortic Valve

SUMMARY:
Collect real-world data on hemodynamic and clinical outcomes of the INSPIRIS RESILIA Aortic Valve, Model 11500A, in subjects requiring replacement of their native or prosthetic aortic valve as the only heart valve procedure during the index procedure, with or without other concomitant procedures.

DETAILED DESCRIPTION:
Subjects in the INDICATE registry study will be enrolled at up to 20 sites in Germany. Up to 500 subjects will be implanted with the INSPIRIS RESILIA Aortic Valve in this registry.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring an aortic valve replacement using the INSPIRIS RESILIA aortic valve according to its intended purpose
2. Patients with standard-of-care pre-procedure imaging evaluation (echocardiography and CT) data available
3. Age ≥ 18 years
4. Provision of written informed consent

Exclusion Criteria:

1. Active endocarditis/myocarditis or endocarditis/myocarditis within 3 months prior to the scheduled aortic valve replacement surgery
2. Emergency procedure
3. Patients requiring a non-aortic heart valve procedure during the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects from Germany who meet all the study inclusion criteria and none of the study exclusion criteria who undergo an aortic valve replacement with the Model 11500A heart valve and voluntary sign a consent form to agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Subject's average mean gradient measurement over time | Prior to discharge (an average of 7 to 10 days after surgery) and at 3 months
  Mean gradient is the average flow of blood through the aortic valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. In general, a higher value is considered worse, and a lower value is considered better but the value is dependent on the size and type of valve.
Subject's average peak gradient measurement over time | Prior to discharge (an average of 7 to 10 days after surgery) and at 3 months
  Peak gradient is the maximum value measured of flow of blood through the aortic valve as measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. In general, a higher valve is considered worse, and a lower value is considered better, but the value is dependent on the size and type of valve.
Amount of aortic transvalvular regurgitation in subjects over time | Prior to discharge (an average of 7 to 10 days after surgery) and at 3 months
  Valvular regurgitation occurs when the valve in the heart does not close tightly allowing some of the blood that was pumped out of the heart to leak back into it. Valvular regurgitation is evaluated by echocardiography over time. It is assessed by four categories, which are "no/trace leak", "a mild leak", "a moderate leak", and "a severe leak". A severe leak indicates a worsening outcome.
Amount of aortic paravalvular regurgitation in subjects over time | Prior to discharge (an average of 7 to 10 days after surgery) and at 3 months
  Paravalvular leak refers to blood flowing through a channel between the implanted artificial valve and the cardiac tissue as a result of inappropriate sealing.
  Paravalvular leak is evaluated by echocardiography over time. It is assessed by four categories, which are "no/trace leak", "a mild leak", "a moderate leak", and "a severe leak". A severe leak indicates a worsening outcome.

SECONDARY OUTCOMES:
Subject's New York Heart Association (NYHA) functional classification at 3 months as compared to baseline. | Baseline and 3 months
  The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Class II. Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Class III. Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV. Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Doenst, Prof. Dr. med., Principal Investigator — Jena University Hospital, University of Jena
Locations (4):
- Germany (4):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Rhön Klinikum Campus Bad Neustadt, Bad Neustadt an der Saale, Bavaria
  - Deutsches Herzzentrum der Charité Berlin, Berlin
  - TUM Klinikum Deutsches Herzzentrum, Munich

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) with other researchers.